CLINICAL TRIAL: NCT06509737
Title: Evaluation of the Effect of Life With Food Allergy Education Based on Pender's Health Promotion Model Given to Parents With Food Allergic Children Face-to-Face and Through Social Media
Brief Title: Evaluation of the Effect of Life With Food Allergy Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ayşe Özeflanili, lecturer, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AnkaraYBU-HEM-AÖZEFLANİLİ
Record Dates: First submitted 2024-07-03; First posted 2024-07-19 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: FOOD ALLERGY; FOOD ALLERGY İN CHİLDREN
Keywords: food allergy; child nursing; child nursing education
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Dependent Variables: The dependent variables of the study are the knowledge scores of the parents in the groups on the Life with Food Allergy Education Data Collection Form.
  Independent Variables: The independent variables of the research are the Food Allergy Life Education application given face to face and via social media, and the sociodemographic characteristics of the child and mother.
  Data Collection Techniques and Tools:Parental Data Collection Form and Life with Food Allergy Education Parent Evaluation Form prepared by the researcher will be used to collect research data.
  The Parent Data Collection Form consists of questions to inquire about the sociodemographic characteristics of the participants, their children's food allergy processes and social media usage characteristics.
  In the study, participants were randomised into two experimental groups. A digital programme was used for block randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOCIAL MEDIA TRAINING INTERVENTION GROUP (Experimental): Life with Food Allergy Training will be held in 3 face-to-face sessions for the 1st intervention group, and the session titles are determined as follows.
  1st Education: Introduction to food allergy, general information 2.Education: Food allergy management, food allergy in school and social environment-use of social support resources 3. Education: Treatment of food allergy, use of adrenaline autoinjectors
  Interventions: Behavioral: social mediagroup
- CLASSİC FACE TO FACE EDUCATİON GROUP (Experimental): Life with food allergy training; The 2nd Intervention Group will share videos created by the trainer with the same training content and visuals as the face-to-face training group on the instagram page to be created on social media. At the same time, it is planned to share posts created from the training content on the actively used page. The participant parents will be ensured to follow the page actively, it will be confirmed that they see the posts by liking them and the follow-up will be done by the researcher.
  Interventions: Behavioral: Face to face group

INTERVENTIONS:
Behavioral: Face to face group — With this research, it is expected that parents' knowledge levels, symptom management levels for food allergies, and treatment knowledge levels will increase by providing Life with Food Allergy Training based on the Health Promotion Model with face-to-face training in parents of children diagnosed with food allergy.
  Other Names: To reveal the changes in the knowledge levels of mothers with children with food allergy through Life with Food Allergy Education
  Arms: CLASSİC FACE TO FACE EDUCATİON GROUP
Behavioral: social mediagroup — With this research, it is expected that parents' knowledge levels, symptom management levels for food allergies, and treatment knowledge levels will increase in parents of children diagnosed with food allergy by providing Life with Food Allergy Education based on the Health Promotion Model through social media.
  Other Names: To reveal the changes in the knowledge levels of mothers with children with food allergy through Life with Food Allergy Education
  Arms: SOCIAL MEDIA TRAINING INTERVENTION GROUP

SUMMARY:
Purpose of the Study It was aimed to reveal the changes in the knowledge levels of mothers with food allergy with Life with Food Allergy Education based on Pender's Health Promotion Model.

With this research, it is expected that there will be an increase in the knowledge levels, symptom management levels for food allergies, and treatment knowledge levels of the parents of children diagnosed with food allergy with Life with Food Allergy Education based on the Health Promotion Model.In the study, one group of subjects, divided into two groups, will be given face-to-face education on life with food allergy. For the other group, online food allergy and life education will be given with the same content via social media.In the study, one group of subjects, divided into two groups, will be given face-to-face education on life with food allergy. For the other group, online food allergy and life education will be given with the same content via social media.

Research Question

1. Is the Life with Food Allergy Training based on Pender's Health Promotion Model given to parents with a child with food allergy effective in increasing the knowledge levels of parents about food allergy?
2. Is there a difference between the knowledge levels of the parents who received the Life with Food Allergy Education Based on Pender's Health Promotion Model given to parents with a child with food allergy face-to-face and through social media? Main Hypotheses of the Study H1: Life with Food Allergy Training based on Pender's Health Promotion Model given to parents with children with food allergy is effective in increasing the knowledge levels of parents about food allergy.

H2: There is a significant difference between the knowledge levels of the parents who received the Life with Food Allergy Education Based on Pender's Health Promotion Model given to parents with children with food allergy face-to-face and through social media.

DETAILED DESCRIPTION:
The aim of this study was to reveal the changes in the knowledge levels of mothers with food allergy through Life with Food Allergy Education based on Pender's Health Promotion Model.

With this research, it is expected to increase the knowledge levels, symptom management levels for food allergies, and treatment knowledge levels of the parents of children diagnosed with food allergy with Life with Food Allergy Education based on the Health Promotion Model.

PURPOSE OF EDUCATION FOR LIFE WITH FOOD ALLERGY 1. Training: General Concepts of Food Allergy Purpose of Training: To ensure that parents have information about food allergy, food allergy symptoms, food allergy diagnosis and treatment process, and anaphylaxis.

Goal of Training: At the end of this training, the parent will

* Knows the definition of food allergy (Question 1).
* Knows what the most common food allergen is (Question 2)
* Knows what the most common and resistant food allergens are (Question 3)
* Knows that medications do not prevent the development of food allergy (4th question)
* Knows what elimination diet is (5th question).
* Knows food allergy diagnostic methods (Question 6).
* Knows not to experiment with food at home during the food allergy treatment process (Question 7)
* Knows that every food can trigger allergies and that different reactions may occur with each encounter. (Questions 8-9)
* Knows the risk factors for food allergy (Question 10).
* Knows what to pay attention to when monitoring food allergy symptoms in babies and children (Question 11).
* Knows the problems that children with severe food allergies may encounter during the treatment process (Question 12)
* He knows to call 112 in case of anaphylaxis (Question 15).
* Knows the foods that most commonly cause food allergies (Question 16).
* Knows the symptoms of food allergy (Question 17).

Training Method:

1st Intervention Group: Web (Social Media) Based Education 2. Intervention Group: Face-to-face Education

Training Material:

1. st Intervention Group: Social media videos - Social media posts
2. nd Intervention Group: Powerpoint presentation - Booklet brochure 2. Training: Food Allergy Process Management Purpose of Training: To provide parents with information about how to manage the food allergy process, what to pay attention to when preparing food, what cross-contamination is, the importance of reading labels, and protecting the child from food allergies outside the home.

Goal of Training: At the end of this training, the parent will

* Knows the importance of reading labels (Questions 18-19)
* Knows what foods are required to be declared on labels in the Regulation in Turkey (Questions 20-22).
* Knows what cross-contamination means and knows what should be taken into consideration to prevent cross-contamination (questions 23-24).
* Knows what to pay attention to when preparing food to prevent contamination (questions 24-28).
* Knows what needs to be done outside the home to protect the child from food allergies (questions 29-30).
* Knows the situations that need to be taken into consideration in the care and nutrition of my child while managing the food allergy process (questions 30-34).
* Knows that the trace amount warning on labels is important. (Question 35)

Training Method:

1. st Intervention Group: Web (Social Media) Based Education
2. nd Intervention Group: Face-to-face Education

Training Material:

1. st Intervention Group: Social media videos - Social media posts
2. nd Intervention Group: Powerpoint presentation - Booklet brochure 3. Training: Treatment of Food Allergy Purpose of Training: To provide parents with information about treatment methods in food allergy, anaphylaxis and anaphylaxis intervention methods, and the use of Penepin.

Goal of Training: At the end of this training, the parent will

* Knows what happens and what to do in case of anaphylaxis (questions 36-37).
* Knows and can count the symptoms of anaphylaxis (Question 38).
* Knows what to pay attention to when prescribing PENEPIN automatic injector (question 39).
* Knows the use of PENEPIN automatic injector (questions 40-43).
* Knows what symptoms to watch for before treating a suspected serious allergic reaction (Question 44).
* Knows that I should always have an emergency action plan and a PENEPIN automatic injector with my child who is at risk of anaphylaxis (Question 45).
* Knows that the prescription and expiration dates of the PENEPIN automatic injector must be followed (Question 46).
* He knows that an anaphylactic reaction may resolve after PENEPIN administration, but symptoms may reoccur after 1-2 hours (Question 48).
* Knows how to obtain reliable information about food allergies (questions 49-50).

Training Method:

1. st Intervention Group: Web (Social Media) Based Education
2. nd Intervention Group: Face-to-face Education

Training Material:

1. st Intervention Group: Social media videos - Social media posts
2. nd Intervention Group: Powerpoint presentation - Booklet brochure

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Face-to-Face Training Group Parent

* The child has a diagnosis of Food Allergy
* Ability to write and speak Turkish
* Volunteering to participate in the research Social Media Education Group İnclusion Criteria
* The child has a diagnosis of Food Allergy
* Ability to write and speak Turkish
* Parent's willingness to participate in the study
* Having a desktop, laptop, tablet or smart phone that can be connected to the internet, actively using social media

Exclusion Criteria:

Face-to-Face Education Group Exclusion Criteria

* The parent has a communication barrier (visual, hearing, diagnosed mental and psychological problems)
* The child has additional chronic diseases other than food allergy
* Parents do not speak Turkish
* Lack of up-to-date telephone information of the family Social Media Education Group Exclusion Criteria
* Parental communication impairment (visual, hearing, diagnosed mental and psychological problems)
* The child has additional chronic diseases other than food allergy
* Parents do not speak Turkish
* Not using social media-internet actively-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
The level of knowledge in mothers before and after receiving education on living with food allergy and the effectiveness of the education will be measured. | From enrollment to the end of treatment at 3 weeks
  Data; It will be collected by the researcher using the Life with Food Allergy Education Parent Evaluation Form, through face-to-face interviews in the face-to-face education group, and through Google Forms in the social media education group. No other scale will be used except the PARENT INFORMATION EVALUATION FORM FORM FOR LIFE TRAINING WITH NUTRIENT ALLERGY BASED ON HEALTH IMPROVEMENT MODEL developed by the author with expert approval. In this scale to be used, an evaluation will be made based on the YES/NO answers to the information questions, which we aim to measure whether the parents know the information in the training content. The scale consists of 50 questions and correct answers will be evaluated over 50 points by giving 1 point for correct answers and 0 points for wrong answers.

CONTACTS AND LOCATIONS:
Overall Officials: AYŞE ÖZEFLANİLİ, Lecturer, Study Chair — Kastamonu University
Locations (2):
- Turkey (Türkiye) (2):
  - Kastamonu Eğitim Araştirma Hastanesi, Kastamonu, Merkez
  - Kastamonu Eğitim Araştirma Hastanesi, Kastamonu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orhan F, Karakas T, Cakir M, Aksoy A, Baki A, Gedik Y. Prevalence of immunoglobulin E-mediated food allergy in 6-9-year-old urban schoolchildren in the eastern Black Sea region of Turkey. Clin Exp Allergy. 2009 Jul;39(7):1027-35. doi: 10.1111/j.1365-2222.2009.03263.x. Epub 2009 Apr 27. PMID 19400894
- See also: Diagnosis and management of food allergy — https://www.cmaj.ca/content/188/15/1087.short
- See also: Motosue MS, Bellolio MF, Van Houten HK, Shah ND, Campbell RL. Increasing emergency department visits for anaphylaxis, 2005-2014. J Allergy Clin Immunol Pract. 2017;5(1):171-175.e3 — https://doi.org/10.1016/j.jaip.2016.08.013
- See also: Sicherer, S. H., Vargas, P. A., Groetch, M. E., Christie, L., Carlisle, S. K., Noone, S., Jones, S.M.. Development and validation of educational materials for food allergy. The Journal of Pediatrics, 2012:160(4), 651-656. — http://doi.org.proxy.lib.fsu.edu/10.1016/j.jpeds.2011.09.056
- See also: National Academies of Sciences, Engineering, and Medicine., Finding a path to safety in food allergy: Assessment of the global burden, causes, prevention, management, and public policy. The National Academies Press,2017. — http://search.ebscohost.com.proxy.lib.fsu.edu/login.aspx?direct=true&db=cat05720a&AN=fsu.PDA002435844&site=eds-live&scope=site
- See also: Kaya, A., Tutar Güven, Ş. ve İşler Dalgıç, A, Sağlığı geliştirme modeline göre verilen eğitimin Türkiye'deki hemşirelik araştırmalarında kullanımı. Hemşirelikte Eğitim ve Araştırma Dergisi, 2018:15, 195-201. — http://jag.journalagent.com

DOCUMENTS (1):
  • Informed Consent Form (2024-08-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT06509737/ICF_000.pdf